CLINICAL TRIAL: NCT03459339
Title: Coordinating Center: Natural History of Barrett's Esophagus Using Tethered Capsule Endomicroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Columbia University (Other); Mayo Clinic (Other); Kansas City Veteran Affairs Medical Center (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, HMS, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-P000604; R01CA184102-01 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-03-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Barrett Esophagus
Keywords: Barrett's Esophagus; Natural History; Capsule; OCT; Tethered Capsule Endomicroscopy
MeSH Terms: conditions — Barrett Esophagus | interventions — Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: 100 participants are enrolled in year 1 in each of five participating centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental OFDI capsule imaging (Experimental): Participants will swallow the OFDI capsule and imaging will be acquired using the OFDI imaging system.
  Intervention: 'Tethered Capsule Endomicroscopy (TCE) Imaging of Barrett's esophagus using OFDI capsule
  Interventions: Device: Tethered Capsule Endomicroscopy (TCE)

INTERVENTIONS:
Device: Tethered Capsule Endomicroscopy (TCE) — Tethered Capsule Endomicroscopy will be used to detect Barrett's Esophagus
  Other Names: OFDI capsule imaging

SUMMARY:
The goal of this research is to follow Barrett's Esophagus participants for 3 years using the tethered capsule endomicroscopy device with distal scanning and a compact imaging system in a multi-site clinical study.

DETAILED DESCRIPTION:
The progression of Barrett's Esophagus will be studied over time using tethered capsule endomicroscopy imaging and will be performed at 5 different clinical centers in the US, namely: Massachusetts General Hospital (MGH),(MA), Mayo Clinic Jacksonville (FL), Mayo Clinic Rochester (MN), Columbia University Medical Center (NY), Kansas City VA Medical Center (MO). MGH will be the coordinating center of this multicenter study. Dr G. Tearney will serve as study Sponsor Investigator.

The purpose of this study is to determine the natural history of Barrett's Esophagus using TCE in participants diagnosed with Barrett's Esophagus and undergoing surveillance endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Participants over the age of 18
* Participants who are capable of giving informed consent
* Participants with a diagnosis of BE without high grade dysplasia, intramucosal adenocarcinoma or esophageal adenocarcinoma, confirmed by endoscopic biopsy
* Participants who had or will have a standard of care EGD within 15 months, exceptions to this can be submitted to the coordinating center (MGH) for approval

Exclusion Criteria:

* Participants with prior endoscopic ablation or resection treatment of BE at enrollment visit
* Participants with esophageal fistula and/or esophageal strictures
* Participants with the inability to swallow capsules
* Concomitant chemotherapy treatment
* Self reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Natural History of Barrett's Esophagus Using Tethered Capsule Endomicroscopy | 4 years
  We will be measuring the size of the area affected by Barrett's.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — MGH
Locations (5):
- United States (5):
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - VA Medical Center, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong J, Grant C, Vuong B, Nishioka N, Gao AH, Beatty M, Baldwin G, Baillargeon A, Bablouzian A, Grahmann P, Bhat N, Ryan E, Barrios A, Giddings S, Ford T, Beaulieu-Ouellet E, Hosseiny SH, Lerman I, Trasischker W, Reddy R, Singh K, Gora M, Hyun D, Queneherve L, Wallace M, Wolfsen H, Sharma P, Wang KK, Leggett CL, Poneros J, Abrams JA, Lightdale C, Leeds S, Rosenberg M, Tearney GJ. Feasibility and Safety of Tethered Capsule Endomicroscopy in Patients With Barrett's Esophagus in a Multi-Center Study. Clin Gastroenterol Hepatol. 2022 Apr;20(4):756-765.e3. doi: 10.1016/j.cgh.2021.02.008. Epub 2021 Feb 4. PMID 33549871